CLINICAL TRIAL: NCT05827809
Title: A Transdiagnostic Psychological Treatment for Anxiety and Depression in Youth: Feasibility, Acceptability and Effect in a Clinical Open Trial in Primary Care
Brief Title: Feasibility, Acceptability and Effect of a Transdiagnostic Psychological Treatment for Anxiety and Depression in Youth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lena Reuterskiold (Other Government)
Responsible Party: Sponsor-Investigator, Lena Reuterskiold, Principal investigator, Region Stockholm
Organization: Region Stockholm (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05939-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Depression; CBT
Keywords: Unified Protocol

STUDY DESIGN:
Intervention Model Description: A clinical open trial evaluating feasibility, acceptability, treatment facilitators as well as treatment effects measured before, after and at 6-month follow-up, for a relatively new transdiagnostic psychological treatment, Unified Protocol, for children and youth with anxiety disorders and/or depression and their parents.
  The therapists in the project will also be in-depth interviewed about the treatment feasibility, compliance and acceptance of the treatment intervention. The study is conducted at 2 primary care clinics with patients and parents seeking for routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol (UP-C/A) for children and youth with anxiety disorders and/or depression (Experimental): A within group design where one clinical manualised intervention, the Unified protocol based on the third-wave of Cognitive Behavior Therapy (CBT), is offered in a 11 session group format to children and adolescents. Parent training is at the same time also offered in a group format. Therapists are trained in the method and receive regular supervision adhering to the evidence-based manual. The group treatment and parent training is delivered face-to- face.
  Interventions: Behavioral: Unified Protocol (UP-C/A) for children and youth with anxiety disorders and /or depression

INTERVENTIONS:
Behavioral: Unified Protocol (UP-C/A) for children and youth with anxiety disorders and /or depression — A transdiagnostic psychological group treatment, Unified Protocol (UP-C/A), one intervention, is tested for children and youth with anxiety disorders and/or depression seeking help in routine care in two primary care locations. Parents are at the same time offered parent training in a group format coupled with the module the children are working on. Feasibility, acceptability and effect of the intervention will be studied, with child self-report, parent-report and therapist assessment.

SUMMARY:
The goal of this open clinical trial is to try out and evaluate a relatively new transdiagnostic psychological treatment, Unified Protocol (UP-C/A), in group format for children and adolescents aged 7-17 years of age with anxiety and/or depression and their parents, in primary care. The therapists in the project will receive training and on-going supervision in UP-C/A.

The main questions it aims to answer are:

1. What are the children's (patients) and parents experience of undergoing a transdiagnostic psychological treatment (UP-C/A) in primary care?
2. What are the therapists' experience of having carried out the treatment with a transdiagnostic psychological treatment (UP-C/A) in primary care?
3. To what extent do children and parents answer self-reports and clinician administered instruments regarding symptoms of anxiety, depression, function and quality of life?
4. To what extent do children and their parents complete the treatment and what is the dropout rate?
5. What does the distribution of diagnoses and co-morbidity look like for patients included in the study?
6. What is the treatment outcome with regard to emotion regulation, symptoms of anxiety, depression, function and quality of life? rated by patients, parents and therapists.
7. To what extent are any effects maintained at a 6-month follow-up?

The participants and their parents will partake in group treatment with Unified Protocol of 11 sessions following an initial screening with the Mini International Neuropsychiatric Interview for children and adolescents (MINI-KID).

DETAILED DESCRIPTION:
Participants in the study are children (7 to 17 years of age) seeking help for anxiety and depression in routine primary care and their parents. The children are screened with the Mini-International Neuropsychiatric Interview for children and adolescents (MINI-KID). Patients assessed as fulfilling criteria for anxiety disorders, obsessive compulsive disorders and/or depression and checked against inclusion and exclusion criteria are informed about the project orally and in writing. Informed consent is obtained verbally and in writing. Recruitment in the two separate clinical sites continues until up to 8 children and their parents constitute a group.

After inclusion children and their parents fill in self-report scales. Some of these self-report scales are already in use in the primary care platform (SDQ) and (R-CADS). The ERICA, KIDSCREEN-10, Client Safisfaction Questionnaire (CSQ) are in paperformat and saved in the clinic. The therapist in the project are asked to fill in a scale that assesses feasibility and acceptability of the intervention, after treatment completion.

Data will be analysed descriptively to answer research question from self-reports from the children, parents and therapist as to satisfaction with treatment, feasibility and acceptability. Treatment effect will be analyzed with paired sample t-test on primary and secondary outcomes.

Therapist have received training in UP-C/A by certified educators in UP and will receive on-going supervision in Unified-Protocol by a UP-certified psychologist, during the group intervention. Also, the group intervention is audio-taped. A random sample of 20% of the sessions will be rated as to compliance with the Unified Protocol. The ratings will be performed by the project investigator, also trained in UP-C/A.

A sample size of about 30 is aimed for based on an average of 6 patients in a group and five treatment groups in total. One clinic is aiming for three groups and the other for two treatment groups. Detailed and clear information about the treatment, time consumption for child and parent groups and a good structure for data collection in the clinics are some planned strategies to minimize dropouts and data loss.

From the overall collected data on child and parent satisfaction, therapist ratings of acceptability, feasibility and treatment effects at a 6-month follow-up, a randomized controlled trial (RCT) is planned for in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17 years of age
* Anxiety syndrome, obsessive-compulsive disorder and/or depression according to the Diagnostic and Statistical Manual of Mental disorders (DSM) as primary problem
* Patients and parents master the Swedish language without interpreter support.
* Willingness/ability to participate after receiving information about what participation entails
* In case of medication, this is on a stable dose, since six weeks

Exclusion Criteria:

* Psychosis, bipolar disorder. substance use syndrome, severely suicidal or pervasive developmental disorder
* Ongoing other psychological treatment
* Abuse or domestic violence

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Emotion Regulation Index for Children and Adolescents (ERICA) | Change from pre intervention to treatment completion at 12 weeks and at a 6 month follow-up.
  A self-report that measures various aspects of emotion regulation with three subscales: 1: Emotional Control (lower scores indicate more emotional control); 2: Emotional Self-Awareness (higher scores indicate more emotional self-awareness); 3: Situational Responsiveness (higher scores indicate more situational responsiveness). 16 items in total. Some scores are reversed. Likert-type scale 1 to 5.

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (R-CADS) | Change from pre intervention to treatment completion at 12 weeks and at a 6 month follow-up.
  A self-report and parent report that measures symptoms of anxiety and depression. Minimum value 0 and maximum 141, where higher scores indicate more anxiety and depression symptoms.
The Strengths and difficulties questionnaire (SDQ) | Change from pre intervention to treatment completion at 12 weeks and at a 6 month follow-up.
  A self-report for children from 11 years of age and their parents that assessing mental health, behavior and peer problems in children 7-17 years. Minimum value 0, maximum 40. Higher scores indicate more problems, apart from the prosocial subscale where higher scores indicate more prosocial behavior.
Kidscreen-10 Index | Change from pre intervention to treatment completion at 12 weeks and at a 6 month follow-up.
  A brief self-report, with 10 items, for children and their parents intended to measure health-related quality of life. Scores range from 1 to 5. Higher scores generally indicate a better quality of life, some scores have to be reversed.
Children's Global Assessment Scale (C-GAS). | Change from pre intervention to treatment completion at 12 weeks and at a 6 month follow-up.
  Assessment of the child´s functional level by the clinician. Scores range from 0-100, with higher scores indicating a higher functioning.
Client Satisfaction Questionnaire (CSQ-8) | After treatment completion at 12 weeks.
  A child and parent self-report on general treatment satisfaction. Scores range from 8-32, with higher scores indicating more satisfaction.
A scale on the Acceptability of Intervention Measure (AIM); Intervention Appropriateness Measure (IAM) and Feasibility of Intervention Measure (FIM). | After the treatment group intervention is completed at 12 weeks.
  Clinician report. Three subscales, with scores ranging from a minimum of 12 and a maximum of 60. Higher scores indicating a better fit with implementation in clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Reuterskiöld, PhD, Principal Investigator — Region Stockholm
Locations (2):
- Sweden (2):
  - Liljeholmens Vårdcentral, Stockholm
  - Älvsjö Vårdcental, Stockholm, Älvsjö